CLINICAL TRIAL: NCT07095751
Title: Pilot Study on Artificial Intelligence-assisted Uro-Cam Catheter Assessment System for Diagnosing Bladder Cancer
Brief Title: Artificial Intelligence-assisted Uro-Cam Catheter Assessment System for Diagnosing Bladder Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Jeremy Yuen Chun TEOH, Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CRE 2025.323
Record Dates: First submitted 2025-07-23; First posted 2025-07-31 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Bladder Cancer
Keywords: AI; Uro-Cam; Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a pilot study investigating the safety, feasibility and diagnostic performance of AI-assisted Uro-Cam catheter assessment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AI Uro-Cam (Experimental): All recruited patients will undergo the AI-assisted Uro-Cam catheter assessment followed by a conventional flexible cystoscopy in the same session. Biopsy will be taken from any suspicious lesion detected upon AI-assisted Uro-Cam catheter assessment or conventional flexible cystoscopy.
  Interventions: Device: AI Uro-Cam

INTERVENTIONS:
Device: AI Uro-Cam — As stated in AI Uro-Cam arm description

SUMMARY:
This is a single-arm study investigating the safety, feasibility and diagnostic performance of AI-assisted Uro-Cam catheter assessment that will be performed at the Prince of Wales Hospital. All patients who are referred to the urology outpatient clinic for hematuria workup, and bladder cancer patients who require follow-up cystoscopy, will be screened for study eligibility. If eligible, patients will be recruited into the study with a proper informed consent. All recruited patients will undergo the AI-assisted Uro-Cam catheter assessment followed by a conventional flexible cystoscopy. The study will be conducted in accordance with the Declaration of Helsinki, and it will be registered in ClinicalTrials.gov.

An AI-assisted Uro-Cam catheter assessment will be arranged for all recruited study subjects. After the AI-assisted Uro- Cam catheter assessment, a conventional flexible cystoscopy will be conducted in the same session. Biopsy will be taken from any suspicious lesion detected upon AI-assisted Uro-Cam catheter assessment or conventional flexible cystoscopy.

After all the procedures, an End-of-study visit will be arranged 4-6 weeks later. The primary outcomes include 30-day complications, and the technical success rate of the AI-assisted Uro-Cam catheter assessment. 30-day complications will be assessed and grading according to the Clavien-Dindo classification. Technical success is defined by the completion of the whole Uro-Cam catheter assessment. The secondary outcomes include the AUC, sensitivity, specificity, positive predictive value, and negative predictive value in detecting histologically confirmed bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above
* Fulfil any one of the following three criteria: (1) Macroscopic haematuria or persistent microscopic haematuria (microscopic haematuria in at least two urine tests), (2) Abnormal urine cytology results (Atypical cells in at least two urine cytology tests, OR Suspicious cells or malignant cells in at least one urine cytology test), (3)History of non-muscle-invasive bladder cancer with complete transurethral resection of bladder tumour performed

Exclusion Criteria:

* Presence of clinically significant cardiovascular disease (History of acute myocardial infarction, presence of uncontrolled angina within 3 months before screening, New York Heart Association Class III or IV congestive heart failure, presence of ventricular arrhythmias, or presence of second-degree or third-degree heart block)
* Any evidence of active urinary tract infection
* Presence of GOLD Stage III or IV chronic obstructive pulmonary disease
* ECOG performance status ≥ 2 (Ambulatory and capable of all self-care but unable to carry our any work activities)
* History of bleeding disorder or use of anti-coagulants
* Presence of other active malignancy
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-31 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
30-day complications | Thirty days after the allocated treatment
  30-day complications will be assessed and grading according to the Clavien-Dindo classification.
Technical success rate | Immediately post-operative
  Technical success is defined by the completion of the whole Uro-Cam catheter assessment.

SECONDARY OUTCOMES:
Performance Evaluation | Thirty days after the allocated treatment
  AUC, sensitivity, specificity, positive predictive value and negative predictive value in detecting bladder cancer will also be evaluated and recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Yuen Chun TEOH, MBBS, FRCSEd, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Britton JP, Dowell AC, Whelan P. Dipstick haematuria and bladder cancer in men over 60: results of a community study. BMJ. 1989 Oct 21;299(6706):1010-2. doi: 10.1136/bmj.299.6706.1010. PMID 2511941
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Vogelmeier CF, Criner GJ, Martinez FJ, Anzueto A, Barnes PJ, Bourbeau J, Celli BR, Chen R, Decramer M, Fabbri LM, Frith P, Halpin DM, Lopez Varela MV, Nishimura M, Roche N, Rodriguez-Roisin R, Sin DD, Singh D, Stockley R, Vestbo J, Wedzicha JA, Agusti A. Global Strategy for the Diagnosis, Management, and Prevention of Chronic Obstructive Lung Disease 2017 Report. GOLD Executive Summary. Am J Respir Crit Care Med. 2017 Mar 1;195(5):557-582. doi: 10.1164/rccm.201701-0218PP. PMID 28128970
- [Background] Hicks KA, Mahaffey KW, Mehran R, Nissen SE, Wiviott SD, Dunn B, Solomon SD, Marler JR, Teerlink JR, Farb A, Morrow DA, Targum SL, Sila CA, Hai MTT, Jaff MR, Joffe HV, Cutlip DE, Desai AS, Lewis EF, Gibson CM, Landray MJ, Lincoff AM, White CJ, Brooks SS, Rosenfield K, Domanski MJ, Lansky AJ, McMurray JJV, Tcheng JE, Steinhubl SR, Burton P, Mauri L, O'Connor CM, Pfeffer MA, Hung HMJ, Stockbridge NL, Chaitman BR, Temple RJ; Standardized Data Collection for Cardiovascular Trials Initiative (SCTI). 2017 Cardiovascular and Stroke Endpoint Definitions for Clinical Trials. Circulation. 2018 Feb 27;137(9):961-972. doi: 10.1161/CIRCULATIONAHA.117.033502. PMID 29483172
- [Background] Hicks KA, Mahaffey KW, Mehran R, Nissen SE, Wiviott SD, Dunn B, Solomon SD, Marler JR, Teerlink JR, Farb A, Morrow DA, Targum SL, Sila CA, Thanh Hai MT, Jaff MR, Joffe HV, Cutlip DE, Desai AS, Lewis EF, Gibson CM, Landray MJ, Lincoff AM, White CJ, Brooks SS, Rosenfield K, Domanski MJ, Lansky AJ, McMurray JJV, Tcheng JE, Steinhubl SR, Burton P, Mauri L, O'Connor CM, Pfeffer MA, Hung HMJ, Stockbridge NL, Chaitman BR, Temple RJ; Standardized Data Collection for Cardiovascular Trials Initiative (SCTI). 2017 Cardiovascular and Stroke Endpoint Definitions for Clinical Trials. J Am Coll Cardiol. 2018 Mar 6;71(9):1021-1034. doi: 10.1016/j.jacc.2017.12.048. PMID 29495982
- [Background] Bray F, Laversanne M, Sung H, Ferlay J, Siegel RL, Soerjomataram I, Jemal A. Global cancer statistics 2022: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2024 May-Jun;74(3):229-263. doi: 10.3322/caac.21834. Epub 2024 Apr 4. PMID 38572751
- [Background] Bastacky S, Ibrahim S, Wilczynski SP, Murphy WM. The accuracy of urinary cytology in daily practice. Cancer. 1999 Jun 25;87(3):118-28. doi: 10.1002/(sici)1097-0142(19990625)87:33.0.co;2-n. PMID 10385442
- [Background] Chan ES, Ng CF, Hou SM, Yip SK. Using urine microscopy and cytology for early detection of bladder cancer in male patients with lower urinary tract symptoms. Int Urol Nephrol. 2011 Jun;43(2):289-94. doi: 10.1007/s11255-010-9856-y. Epub 2010 Nov 4. PMID 21053072
- [Background] Sharp VJ, Barnes KT, Erickson BA. Assessment of asymptomatic microscopic hematuria in adults. Am Fam Physician. 2013 Dec 1;88(11):747-54. PMID 24364522
- [Background] Ritchie CD, Bevan EA, Collier SJ. Importance of occult haematuria found at screening. Br Med J (Clin Res Ed). 1986 Mar 8;292(6521):681-3. doi: 10.1136/bmj.292.6521.681. PMID 3081223
- [Background] Babjuk M, Burger M, Capoun O, Cohen D, Comperat EM, Dominguez Escrig JL, Gontero P, Liedberg F, Masson-Lecomte A, Mostafid AH, Palou J, van Rhijn BWG, Roupret M, Shariat SF, Seisen T, Soukup V, Sylvester RJ. European Association of Urology Guidelines on Non-muscle-invasive Bladder Cancer (Ta, T1, and Carcinoma in Situ). Eur Urol. 2022 Jan;81(1):75-94. doi: 10.1016/j.eururo.2021.08.010. Epub 2021 Sep 10. PMID 34511303
- [Background] Peterson LM, Reed HS. Hematuria. Prim Care. 2019 Jun;46(2):265-273. doi: 10.1016/j.pop.2019.02.008. Epub 2019 Apr 1. PMID 31030828
- [Background] Roth V, Espino-Grosso P, Henriksen CH, Canales BK. Office Cystoscopy Urinary Tract Infection Rate and Cost before and after Implementing New Handling and Storage Practices. Urol Pract. 2021 Jan;8(1):23-29. doi: 10.1097/UPJ.0000000000000162. Epub 2020 May 27. PMID 37145433
- [Background] Khadhouri S, Gallagher KM, MacKenzie KR, Shah TT, Gao C, Moore S, Zimmermann EF, Edison E, Jefferies M, Nambiar A, Mannas MP, Lee T, Marra G, Lillaz B, Gomez Rivas J, Olivier J, Assmus MA, Ucar T, Claps F, Boltri M, Burnhope T, Nkwam N, Tanasescu G, Boxall NE, Downey AP, Lal AA, Anton-Juanilla M, Clarke H, Lau DHW, Gillams K, Crockett M, Nielsen M, Takwoingi Y, Chuchu N, O'Rourke J, MacLennan G, McGrath JS, Kasivisvanathan V; IDENTIFY Study group. The IDENTIFY study: the investigation and detection of urological neoplasia in patients referred with suspected urinary tract cancer - a multicentre observational study. BJU Int. 2021 Oct;128(4):440-450. doi: 10.1111/bju.15483. Epub 2021 Sep 8. PMID 33991045
- [Background] O'Connor E, McVey A, Demkiw S, Lawrentschuk N, Murphy DG. Assessment and management of haematuria in the general practice setting. Aust J Gen Pract. 2021 Jul;50(7):467-471. doi: 10.31128/AJGP-03-21-5892. PMID 34189542
- [Background] Matulewicz RS, Meeks JJ. Blood in the Urine (Hematuria). JAMA. 2016 Oct 11;316(14):1508. doi: 10.1001/jama.2016.4716. No abstract available. PMID 27727385